CLINICAL TRIAL: NCT01117155
Title: A Pilot Study Evaluating 18F-L-Thymidine (FLT) PET Imaging in Children With Gliomas
Status: Withdrawn | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 100105; 10-C-0105
Record Dates: First submitted 2010-05-04; First posted 2010-05-05 (Estimated); Last update posted 2019-12-12 (Actual); Status verified 2012-10-22

CONDITIONS: Ependymoma; Brainstem Glioma; Astrocytoma; Glioblastoma Multiforme; PNET
Keywords: Brain Tumor; Imaging; FLT; FDG; Spectroscopy; Glioma; Glioblastoma Multiforme; Astrocytoma
MeSH Terms: conditions — Ependymoma; Astrocytoma; Glioblastoma; Neuroectodermal Tumors, Primitive; Brain Neoplasms; Glioma

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Background:

* Children with brain tumors often have magnetic resonance imaging (MRI) scans to see if the tumor has responded to therapy or to see if the tumor has grown. Sometimes, it is difficult to tell if the scan is abnormal because of tumor size or shape, swelling, scar tissue, or dead tissue. Because brain tumor biopsies require surgery, researchers are looking for more noninvasive ways of evaluating brain tumors.
* Positron emission tomography (PET) scans use a radioactive sugar known as 18F-FDG to try to determine if a tumor is active or not. Active tumors generally take up more sugar than the surrounding tissue, but because normal brain tissue uses the same sugar as brain tumors, it is then difficult to tell if tumor tissue is taking up sugar or not. A different radioactive agent, 18F-FLT, is now being studied in some adults with different kinds of tumors. Researchers are interested in determining whether it is possible to use this agent as a marker of tumor activity in children.

Objectives:

* To determine the safety and effectiveness of 18F-FLT for pediatric glioma scans.
* To compare the results of 18F-FLT studies with studies using the radioactive agents 18F-FDG and 1H-MRSI.

Eligibility:

- Children less than 18 years of age who are having radiation therapy to treat malignant gliomas.

Design:

* Participants will have scanning tests before radiation therapy, 1 to 3 weeks after radiation therapy, and if researchers suspect that the tumor is growing.
* This study will involve three separate imaging tests (1H-MRSI, 18F-FDG PET, and 18F-FLT PET).
* Proton spectroscopy (1H-MRSI) is a procedure that is similar to MRI and is performed in the same scanner as an MRI. Because this scan is long (2-3 hours), most children will receive medications from an anesthesiologist so that they can sleep through the procedure.
* Within 2 weeks of the 1H-MRSI scan, participants will have the PET scans with both the standard contrast agent (18F-FDG) and the experimental agent (18F-FLT). These scans will last approximately 1 hour each.

DETAILED DESCRIPTION:
BACKGROUND:

* A limitation of current investigational therapy for patients with brain tumors is assessment of response.
* (18)F-FDG PET is commonly used to assess tumor metabolism. However, normal brain uses glucose as an energy source, resulting in increased background FDG uptake, which confounds results and makes it difficult to distinguish normal from neoplastic activity.
* Newer imaging techniques that noninvasively assess metabolic and physiologic characteristics of brain tumor tissue are being developed to identify biomarkers of clinical efficacy in trials of new molecularly targeted agents.
* (18)F-fluorothymidine (FLT) is a PET radiopharmaceutical that is taken up by proliferating cells and may therefore serve as a surrogate marker of early response or lack of response to treatment.
* This study will prospectively evaluate (18)F-FLT in children undergoing radiation therapy for gliomas.

OBJECTIVES:

Primary objectives:

* Determine the feasibility of (18)F-FLT PET imaging in pediatric patients with malignant gliomas
* Determine the ability of (18)F-FLT PET imaging to detect treatment changes in pediatric patients with malignant gliomas undergoing radiation therapy

Secondary objectives:

* Determine the safety and toxicity profile of PET imaging using (18)F-FLT in pediatric patients with malignant gliomas
* To correlate changes in (18)F-FLT PET before and after radiation with outcome (12 month PFS)
* To compare the performance of (18)F-FLT-PET to that of MR perfusion, proton magnetic resonance spectroscopy (1H-MRSI) and (18)F-FDG PET in prediction of tumor response, time to progression and overall survival time.

ELIGIBILITY:

* Children less than 18 years of age with malignant gliomas for whom radiation therapy is prescribed.
* Adequate organ function defined as:

  * Hepatic: SGOT, SGPT less than 5 times the ULN; total and direct bilirubin less than or equal to 2 times the ULN
  * Renal: Serum creatinine must be within the upper limit of normal values
* Fasting serum glucose less than 150 mg/dL
* Negative serum or urine pregnancy test in females of childbearing potential

DESIGN:

-Patients will undergo MRI (with 1H-MRSI and perfusion), (18)F-FLT PET and (18)F-FDG PET within 2 weeks of each other at the following time points: pre-radiation therapy, 1-3 weeks post-radiation therapy, and at the time of suspected progression.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Age: 1 year to less than 18 years of age
* Diagnosis: Patients must have a histologic diagnosis of a malignant glioma for which radiation therapy is prescribed. Patients with DIPG or optic pathway gliomas are exempt from this requirement and do not require a histologic diagnosis. All patients must have evaluable (not necessarily measurable) disease.
* Weight less than or equal to 70 kg (to limit radioisotope exposure to maximum adult dose)
* All patients or their legal guardians must sign a document of informed consent indicating their awareness of the investigational nature and risks of this study.
* Organ Function: Patients must have adequate organ function defined as:

Hepatic: SGOT/AST, SGPT/ALT less than 5 times the ULN, Total bilirubin less than or equal to 2 times the ULN

Renal: Serum creatinine within the upper limit of normal values for age

Serum Glucose: less than 150 mg/dL

* Female patients of childbearing potential must have a negative serum or urine pregnancy test
* Patients must be able to undergo both the FLT and FDG PET without the use of general anesthesia.

EXCLUSION CRITERIA:

* Patients unable to undergo MR imaging for any reason (including but not limited to the presence of a metallic implant that is not MRI compatible)
* Pregnant women are excluded because of known harmful effects of radiation on the fetus and the unknown effects of strong magnetic fields and Gadolinium contrast agents on the fetus.
* Any patient with a history of severe reaction (requiring medication) to Gd-DTPA, FDG or FLT.
* Any patient with permanent dental hardware, which, in the judgment of the Principal Investigator, would interfere with obtaining spectroscopy in the area of the tumor.
* Any patient who has begun an investigational agent within 48 hours prior to receiving (18)F-FLT.

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2010-04-23; Study Completion 2012-10-22

CONTACTS AND LOCATIONS:
Overall Officials: Katherine E Warren, M.D., Principal Investigator — National Cancer Institute (NCI)

REFERENCES:
- [Background] Rekate HL, Rakfal SM. Low-grade astrocytomas of childhood. Neurol Clin. 1991 May;9(2):423-40. PMID 1944108
- [Background] Therasse P, Arbuck SG, Eisenhauer EA, Wanders J, Kaplan RS, Rubinstein L, Verweij J, Van Glabbeke M, van Oosterom AT, Christian MC, Gwyther SG. New guidelines to evaluate the response to treatment in solid tumors. European Organization for Research and Treatment of Cancer, National Cancer Institute of the United States, National Cancer Institute of Canada. J Natl Cancer Inst. 2000 Feb 2;92(3):205-16. doi: 10.1093/jnci/92.3.205. PMID 10655437
- [Background] Gururangan S, Cavazos CM, Ashley D, Herndon JE 2nd, Bruggers CS, Moghrabi A, Scarcella DL, Watral M, Tourt-Uhlig S, Reardon D, Friedman HS. Phase II study of carboplatin in children with progressive low-grade gliomas. J Clin Oncol. 2002 Jul 1;20(13):2951-8. doi: 10.1200/JCO.2002.12.008. PMID 12089224